CLINICAL TRIAL: NCT02528981
Title: Effect of Probiotics on GBS Colonization Status During Pregnancy: A Pilot Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Collaborators: Chr Hansen (Industry)
Responsible Party: Principal Investigator, Mary Sharpe, Associate Professor, Toronto Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: REB 2012-165
Record Dates: First submitted 2015-08-18; First posted 2015-08-19 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Group B Streptococcal Infection
Keywords: GBS; Probiotics; Group B Streptococcal; Pregnancy
MeSH Terms: conditions — Streptococcal Infections | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Experimental): L. rhamnosus GR-1 and L. reuteri RC-14 will be supplied to 100 randomized pregnant people in gelatin capsules containing 2.5 billion viable cells of each strain (CFU). These organisms have been previously shown to colonize the vagina after being taken orally (11) and displace the pathogens causing bacterial vaginosis (12) and vaginal yeast infections (13), and have been shown to be an effective treatment, or accessory to treatment of these conditions. (7- 9, 13)
  Interventions: Drug: Probiotic
- Placebo (Placebo Comparator): Placebo capsules will be supplied to 100 randomized pregnant people in gelatin capsules that are identical to the probiotics that the experimental group will receive.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Probiotic — Lactobacillus GR-1 and RC-14
  Arms: Probiotic
Drug: Placebo
  Arms: Placebo

SUMMARY:
Group B Streptococcus (GBS) is the leading cause of neonatal morbidity and mortality in Canada. It may be passed from a study participant colonized in the genital tract by GBS to their baby during vaginal birth. While approximately 10 to 30% of pregnant people harbour GBS in the vagina or rectum, the incidence of neonatal GBS disease is 1 to 2 infants per 1000 births. The use of intrapartum antibiotics to treat colonized individuals with or without risk factors has led to a 70% decline in the incidence of early-onset GBS sepsis in the past decade. Despite this impressive decline, antibiotic resistance has become a major public health concern. Association between intrapartum antibiotic use and ampicillin resistance in E. coli isolated from neonates has previously been documented. Furthermore, while GBS has remained sensitive to penicillin, 20% are resistant to erythromycin and clindamycin, which are alternate drugs for patients allergic to penicillin. Alternative approaches are therefore needed to reduce the risk of GBS infection.

We therefore propose to study the use of Lactobacillus rhamnosus GR-1 and Lactobacillus reuteri RC-14 (Lactobacillus fermentum RC-14) in the colonization status of GBS in pregnant people. Lactobacilli are part of normal gut and vaginal flora and have been widely used as probiotics to treat various conditions. In particular, these two strains have shown to be beneficial in the treatment of urinary tract infections and bacterial vaginosis. Our study design involves recruiting two hundred pregnant people (one hundred in each arm) through various midwifery practices in the GTA at the end of their first trimester of pregnancy. These individuals will be randomized to receive probiotics or placebo for twelve weeks of their pregnancies and will be cultured before delivery to determine their colonization status. The capsules with probiotics and placebo will be provided free of charge. The study design was chosen to minimize the cost and clients' visits to the clinic as vaginal/rectal swabs are routinely offered at 35-37 weeks of gestation.

DETAILED DESCRIPTION:
Study Abstract

Group B Streptococcus (GBS) is the leading cause of neonatal morbidity and mortality in Canada. It may be passed from a study participant colonized in the genital tract by GBS to their baby during vaginal birth. While approximately 10 to 30% of pregnant people harbour GBS in the vagina or rectum, the incidence of neonatal GBS disease is 1 to 2 infants per 1000 births. The use of intrapartum antibiotics to treat colonized individuals with or without risk factors has led to a 70% decline in the incidence of early-onset GBS sepsis in the past decade. Despite this impressive decline, antibiotic resistance has become a major public health concern. Association between intrapartum antibiotic use and ampicillin resistance in E. coli isolated from neonates has previously been documented. Furthermore, while GBS has remained sensitive to penicillin, 20% are resistant to erythromycin and clindamycin, which are alternate drugs for patients allergic to penicillin. Alternative approaches are therefore needed to reduce the risk of GBS infection.

We therefore propose to study the use of Lactobacillus rhamnosus GR-1 and Lactobacillus reuteri RC-14 (Lactobacillus fermentum RC-14) in the colonization status of GBS in pregnant people. Lactobacilli are part of normal gut and vaginal flora and have been widely used as probiotics to treat various conditions. In particular, these two strains have shown to be beneficial in the treatment of urinary tract infections and bacterial vaginosis. Our study design involves recruiting two hundred pregnant people (one hundred in each arm) through various midwifery practices in the GTA at the end of their first trimester of pregnancy. These individuals will be randomized to receive probiotics or placebo for twelve weeks of their pregnancies and will be cultured before delivery to determine their colonization status. The capsules with probiotics and placebo will be provided free of charge. The study design was chosen to minimize the cost and clients' visits to the clinic as vaginal/rectal swabs are routinely offered at 35-37 weeks of gestation.

As lactobacilli are part of the human gut flora and have low pathogenicity, no adverse reaction to lactobacilli or placebo is anticipated, though some clients may experience flatulence. The process of reporting unexpected or adverse events is outlined in the Case Report Form (CRF). Concerns relating to the integration of this study into the practices of midwives in the community will be mitigated by letters of information to midwives and clients, informed choice discussions between the researchers and study participants, and letters of consent.

Background

Group B Streptococcus (GBS) is a gram-positive bacterium. The gut is the bodily reservoir for GBS, and the most likely source of vaginal colonization. While part of the normal vaginal flora and usually of no noticeable consequence to people, GBS emerged in the 1970s as the leading cause of neonatal morbidity and mortality. A primary risk factor for neonatal contraction is colonization of the carrier's vaginal tract, with the bacteria being passed to the baby as it travels through the birth canal, or by being spread to the amniotic fluid. This vertical transmission can lead to early-onset GBS disease of the newborn (EOGBSD), which manifests in the first 7 days of life, and can be fatal. Therefore, current clinical recommendations focus on the prevention of GBS-associated diseases by monitoring and managing the GBS colonization status of the pregnant person in an attempt to reduce the probability of the neonate contracting a GBS infection during birth. Currently, midwives in Ontario are advised to offer all clients culture screening for GBS at 35-37 weeks gestation. People who screen positive for GBS are to be offered intrapartum antibiotic prophylaxis (IAP) either universally, or based on other risk factors. IAP is not specifically recommended for who can reasonably be expected to be GBS-free (i.e. screened negative for GBS when tested at 35-37 weeks).

While EOGBSD is potentially very serious, the use of IAP is associated with its own risks. Concomitant with the use of IAP are the risks of: maternal anaphylaxis, emergence of antibiotic-resistant strains of bacteria, infection with non-GBS organisms, colonization with yeast, the development of allergies and asthma. In addition, because IAP requires clients to labour attached to an IV at various time-points throughout their labour, IAP is a disruption to the natural course of labour and delivery that midwives try to facilitate. Furthermore, GBS screening and positive status can be very stressful for people. Therefore, in an attempt to eliminate stress, the need for IAP and the risks and inconvenience associated with it, midwives offer certain strategies to clients in an attempt to reduce the probability that they will screen positive for the GBS bacteria. Homeopathy, garlic suppositories, and probiotic capsules are all methods midwives and their clients use in an attempt to prevent vaginal colonization by GBS. However, there is no evidence to support or refute the use of these remedies.

Probiotics are defined as viable microbial food supplements which, if given in adequate quantities, confer a health benefit to the host. Bacteria of the lactobacillus sp. are the most common in probiotic capsule preparations, and they are also the most common type of organism found in the natural vaginal flora. The natural vaginal flora play an important role in dislodging and inhibiting pathogens. The rationale for the use of probiotics then, is the return of the vaginal flora to their healthy, natural state. Indeed, probiotics have been shown to alter the vaginal flora being an effective supplement in the treatment and cure of bacterial vaginosis, and vulvovaginal yeast infections. Probiotic capsules are considered safe for use in pregnancy.

Research Question

Does taking probiotics for 12 weeks during pregnancy effect the GBS colonization status of people at 35-37 weeks of pregnancy?

Study Design

Probiotic Capsules

L. rhamnosus GR-1 and L. reuteri RC-14 will be supplied to pregnant people in gelatin capsules containing 2.5 billion viable cells of each strain (CFU). These organisms have been previously shown to colonize the vagina after being taken orally and displace the pathogens causing bacterial vaginosis and vaginal yeast infections, and have been shown to be an effective treatment, or accessory to treatment of these conditions. This formulation has been previously approved for use in clinical trials in Canada. The probiotics and placebo are provided in gelatin capsules. The use of gelatin capsules may be prohibitive for some individuals who are vegetarian, vegan, Muslim or Jewish.

Subjects & Randomization

This is a randomized, placebo-controlled trial. In order to achieve 80% statistical power and a p value of 0.05 with the assumption that 20% of people in the placebo group will become GBS positive, 200 clients will be recruited from participating midwifery clinics in the Greater Toronto Area and randomized into each study arm (2 groups of 100). Clients will be offered entry to the study upon beginning midwifery care, and will be provided with either oral Lactobacillus GR-1 and RC-14 or placebo (cellulose, magnesium stearate). Two capsules are to be taken once daily for 12 weeks from 24 weeks of pregnancy until their GBS swab test which is taken at 35-37 weeks of pregnancy, routine to the standard of midwifery care.

Relevance

The hope is that this study will shed some light on the utility of probiotics in midwifery care as pertaining to GBS colonization. This study may provide evidence that probiotic prophylaxis is an effective, low-risk strategy that we can continue to offer to clients to reduce their risk of GBS colonization and thus, the need for IAP and the risks and inconvenience associated with it. Alternatively, this study will provide evidence that probiotics are not an efficacious supplement to offer, and should not be recommended, as the capsules are quite costly and their purchase, or the decision-making process around whether they can or should obtain capsules, may place undue hardship on some people.

Safety and Adverse Event Monitoring

It is the investigators mandate to protect the safety of the study participants. The possibility of adverse events through the use of placebo and probiotics is extremely minimal. Participants are informed that there is a small chance of experiencing flatulence with the capsules. Any unexpected or adverse events will be reported immediately by participants to their midwife, who will document it on the Case Report Form (CRF) and will notify the Practice Research Collaborator (PRC) at their clinic. The PRC then would notify the PI or their delegate for further investigation. As study participants are all in the direct care of midwives who are aware of the study and their client's participation in the study, midwives will manage, consult, or transfer care according to their College guidelines in the event of an unexpected or adverse event. The PRC and PI or their delegates are responsible for documenting any AEs in the CRF. The PI, in collaboration with the QI and Co-I, where applicable, will determine the severity of the AE and causality. Severe AEs are reportable to the REB and Health Canada. Study participants who experience unexpected, adverse, or severe adverse events will be considered for exclusion from the study.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant prior to 23 weeks' gestation
* Singleton pregnancy
* Greater than 18 years of age
* Lesser than 45 years of age
* Signed Informed Consent
* Consent to GBS swab that will be offered at the 35-37 week visit
* Consent to chart review at study conclusion

Exclusion Criteria:

* Multifetal pregnancy
* Fetal complications
* History of preterm birth/second trimester loss
* Significant maternal medical complications
* Unable to provide informed consent
* 18 years of age or lesser than 18 years of age
* 45 years of age or greater than 45 years of age
* HIV positive
* Immuno-compromised E.g.: Persons with AIDS; cancer and transplant patients who are taking certain immunosuppressive drugs; and those with inherited diseases that affect the immune system (e.g., congenital agammaglobulinemia, congenital IgA deficiency).
* History of previous child affected by Early Onset GBS Disease (EOGBSD)
* GBS bacteruria in pregnancy
* Antibiotic treatment required during study period
* Enrolled in other research with a drug
* Taking another probiotic supplement

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2015-08; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
The GBS colonization status of people as determined by a vaginal/rectal swab | After 12 weeks of taking capsules
  The primary outcome of this study is the GBS colonization status of people as determined by a vaginal/rectal swab, routine to the standard course of midwifery care, taken at 35-37 weeks of pregnancy. Thus, clients are asked to participate in the study for approximately 12 weeks, as per the course of probiotic/placebo. Clients will stop taking the capsules after 12 weeks and once the swab has been performed

CONTACTS AND LOCATIONS:
Overall Officials: Mary Sharpe, PhD, Principal Investigator — Toronto Metropolitan University
Locations (1):
- Ryerson University, Toronto, Ontario, Canada

REFERENCES:
- [Background] Stoll BJ, Hansen NI, Sanchez PJ, Faix RG, Poindexter BB, Van Meurs KP, Bizzarro MJ, Goldberg RN, Frantz ID 3rd, Hale EC, Shankaran S, Kennedy K, Carlo WA, Watterberg KL, Bell EF, Walsh MC, Schibler K, Laptook AR, Shane AL, Schrag SJ, Das A, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Early onset neonatal sepsis: the burden of group B Streptococcal and E. coli disease continues. Pediatrics. 2011 May;127(5):817-26. doi: 10.1542/peds.2010-2217. Epub 2011 Apr 25. PMID 21518717
- [Background] Verani JR, McGee L, Schrag SJ; Division of Bacterial Diseases, National Center for Immunization and Respiratory Diseases, Centers for Disease Control and Prevention (CDC). Prevention of perinatal group B streptococcal disease--revised guidelines from CDC, 2010. MMWR Recomm Rep. 2010 Nov 19;59(RR-10):1-36. PMID 21088663
- [Background] Darling E, Saurette K. Clinical Practice Guideline No.11: Group B Streptococcus: Prevention and Management in Labour. Toronto: Association of Ontario Midwives 2010.
- [Background] Money DM, Dobson S; Canadian Paediatric Society, Infectious Diseases Commitee. RETIRED: The prevention of early-onset neonatal group B streptococcal disease. J Obstet Gynaecol Can. 2004 Sep;26(9):826-40. doi: 10.1016/s1701-2163(16)30157-8. English, French. PMID 15361281
- [Background] Kalliomaki M, Salminen S, Isolauri E. Positive interactions with the microbiota: probiotics. Adv Exp Med Biol. 2008;635:57-66. doi: 10.1007/978-0-387-09550-9_5. PMID 18841703
- [Background] Reid G, Dols J, Miller W. Targeting the vaginal microbiota with probiotics as a means to counteract infections. Curr Opin Clin Nutr Metab Care. 2009 Nov;12(6):583-7. doi: 10.1097/MCO.0b013e328331b611. PMID 19741517
- [Background] Anukam K, Osazuwa E, Ahonkhai I, Ngwu M, Osemene G, Bruce AW, Reid G. Augmentation of antimicrobial metronidazole therapy of bacterial vaginosis with oral probiotic Lactobacillus rhamnosus GR-1 and Lactobacillus reuteri RC-14: randomized, double-blind, placebo controlled trial. Microbes Infect. 2006 May;8(6):1450-4. doi: 10.1016/j.micinf.2006.01.003. Epub 2006 Mar 29. PMID 16697231
- [Background] Martinez RC, Franceschini SA, Patta MC, Quintana SM, Gomes BC, De Martinis EC, Reid G. Improved cure of bacterial vaginosis with single dose of tinidazole (2 g), Lactobacillus rhamnosus GR-1, and Lactobacillus reuteri RC-14: a randomized, double-blind, placebo-controlled trial. Can J Microbiol. 2009 Feb;55(2):133-8. doi: 10.1139/w08-102. PMID 19295645
- [Background] Martinez RC, Franceschini SA, Patta MC, Quintana SM, Candido RC, Ferreira JC, De Martinis EC, Reid G. Improved treatment of vulvovaginal candidiasis with fluconazole plus probiotic Lactobacillus rhamnosus GR-1 and Lactobacillus reuteri RC-14. Lett Appl Microbiol. 2009 Mar;48(3):269-74. doi: 10.1111/j.1472-765X.2008.02477.x. Epub 2009 Feb 2. PMID 19187507
- [Background] Reid G, Kirjaivanen P. Taking probiotics during pregnancy. Are they useful therapy for mothers and newborns? Can Fam Physician. 2005 Nov;51(11):1477-9. PMID 16353828
- [Background] Morelli L, Zonenenschain D, Del Piano M, Cognein P. Utilization of the intestinal tract as a delivery system for urogenital probiotics. J Clin Gastroenterol. 2004 Jul;38(6 Suppl):S107-10. doi: 10.1097/01.mcg.0000128938.32835.98. PMID 15220672
- [Background] Burton JP, Cadieux PA, Reid G. Improved understanding of the bacterial vaginal microbiota of women before and after probiotic instillation. Appl Environ Microbiol. 2003 Jan;69(1):97-101. doi: 10.1128/AEM.69.1.97-101.2003. PMID 12513982
- [Background] Reid G, Beuerman D, Heinemann C, Bruce AW. Probiotic Lactobacillus dose required to restore and maintain a normal vaginal flora. FEMS Immunol Med Microbiol. 2001 Dec;32(1):37-41. doi: 10.1111/j.1574-695X.2001.tb00531.x. PMID 11750220
- [Background] Bocking A. Probiotic therapy for the reversal of Bacterial Vaginosis in pregnancy (ProVIP). ClinicalTrials.gov [Internet]. Accessed January 2013. Available from: http://www.clinicaltrials.gov/ct2/show/NCT01697683?term=Bocking%2C+A&rank=10
- [Background] Reid G. Effects of probiotics on rheumatoid arthritis patients. ClinicalTrials.gov [Internet]. Accessed January 2013. Available from: http://www.clinicaltrials.gov/ct2/show/NCT00664820?term=%22Canada%22+AND+%22Probiotics%22&rank=2